CLINICAL TRIAL: NCT01356160
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Response Guided Therapy With GS-5885 Alone or in Combination With GS-9451 With Peginterferon Alfa 2a and Ribavirin in Treatment Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection
Brief Title: GS-5885 Alone or in Combination With GS-9451 With Peginterferon Alfa 2a and Ribavirin in Treatment Chronic Genotype 1 Hepatitis C Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-256-0148
Record Dates: First submitted 2011-05-02; First posted 2011-05-19 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy HCV RNA; Protease inhibitor; Treatment naïve; GS-5885; GS-9451
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ledipasvir; GS-9451; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Active Comparator): RGT with GS-5885 30 mg QD + GS-9451 200 mg QD + PEG/RBV
  Interventions: Drug: GS-5885; Drug: GS-9451; Biological: peginterferon alfa-2a; Drug: ribavirin tablet
- Arm 2 (Placebo Comparator): RGT with GS-5885 30 mg QD + GS-9451 placebo QD + PEG/RBV
  Interventions: Drug: GS-5885; Biological: peginterferon alfa-2a; Drug: ribavirin tablet; Drug: GS-9451 Placebo

INTERVENTIONS:
Drug: GS-5885 — tablet, 30 mg QD
Drug: GS-9451 — tablet, 200 mg QD
  Arms: Arm 1
Biological: peginterferon alfa-2a — (solution for injection) 180 µg/week
Drug: ribavirin tablet — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID)
Drug: GS-9451 Placebo — Placebo to match GS-9451 QD
  Arms: Arm 2

SUMMARY:
This is a Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Response Guided Therapy with GS-5885 Alone or in Combination with GS-9451 with Peginterferon Alfa 2a and Ribavirin in Treatment Naïve Subjects with Chronic Genotype 1 Hepatitis C Virus Infection.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-70 years of age
* Chronic HCV infection
* Subjects must have liver biopsy results (≤ 2 years prior to Screening) indicating the absence of cirrhosis.
* Monoinfection with HCV genotype 1
* HCV RNA > 10^4 IU/mL at Screening
* HCV treatment naïve
* Candidate for PEG/RBV therapy
* Body mass index (BMI) 18-36 kg/m2, inclusive
* Agree to use two forms of highly effective contraception methods for the duration of the study and for 7 months after the last dose of study medication. Females of childbearing potential must have negative pregnancy test at Screening and Baseline.

Exclusion Criteria:

* Pregnant female or male with pregnant female partner
* Exceed defined thresholds for leukopenia, neutropenia, anemia, thrombocytopenia, thyroid stimulating hormone (TSH)
* Diagnosis of autoimmune disease, decompensated liver disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), HIV, hepatitis B virus (HBV), hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers), hemoglobinopathy, retinal disease, or are immunosuppressed.
* Subjects with current use of amphetamines, cocaine, opiates (e.g., morphine, heroin), or ongoing alcohol abuse are excluded. Patients on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to Screening may be included into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the antiviral efficacy of response guided therapy. | Through 24 weeks post-treatment
  To evaluate the antiviral efficacy as measured by sustained virologic response (SVR, defined as plasma HCV RNA < Lower Limit of Quantification (LLoQ) at 24 weeks post-treatment) of response guided therapy (RGT) with GS-5885 + GS-9451 + PEG/RBV, or GS-5885 + PEG/RBV.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of each regimen. | Through 24 weeks post-treatment
  The primary safety endpoint is any AE leading to permanent discontinuation of study drugs.
To characterize viral dynamics of GS-5885 and GS-9451 when administered with PEG and RBV. | Through Day 10 on study
  HCV RNA levels, pharmacokinetics and viral sequencing
To characterize the viral resistance to GS-5885 and GS-9451 when administered in combination with PEG and RBV. | 12 or 24 weeks
  Plasma samples will be collected and stored at each visit for possible resistance analysis.
To characterize steady state pharmacokinetics of GS-5885 and GS-9451 when administered with PEG and RBV. | Through 48 weeks of treatment
  Plasma concentrations of the study drug over time will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Chair — Gilead Sciences
Locations (22):
- United States (20):
  - Tucson, Arizona
  - Beverly Hills, California
  - Coronado, California
  - Costa Mesa, California
  - San Diego, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Bradenton, Florida
  - Baltimore, Maryland
  - Burlington, Massachusetts
  - Kansas City, Missouri
  - Forest Hills, New York
  - Manhasset, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
- Herston, Queensland, Australia
- San Juan, Puerto Rico